CLINICAL TRIAL: NCT01088802
Title: A Phase II Study on Treatment De-Intensification in Favorable Squamous Cell Carcinoma of the Oropharynx
Brief Title: Treatment De-Intensification for Squamous Cell Carcinoma of the Oropharynx
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J0988; NA_00026771 (Other: JHM IRB)
Record Dates: First submitted 2009-08-04; First posted 2010-03-17 (Estimated); Results first posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Squamous Cell Carcinoma of Oropharynx
Keywords: Squamous Cell Carcinoma; Oropharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose de-escalating radiation therapy with chemotherapy (Experimental): This protocol combines selective radiation therapy dose de-escalation (from 70 Gy to 63 Gy and from 58.1 Gy to 50.75 Gy, same number of fractions (N=35) in 7 weeks) in patients with HPV-associated cancers of the oropharynx
  Interventions: Radiation: IMRT; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Radiation: IMRT — Dose de-escalation (from 70 Gy to 63 Gy and from 58.1 Gy to 50.75 Gy, same number of fractions (N=35) in 7 weeks)
Drug: Cisplatin — Cisplatin will be administered weekly for the first 3 weeks and the last 3 weeks of radiation. Patients will not receive chemotherapy during week 4 of treatment.
Drug: Carboplatin — Carboplatin will be administered weekly during the 7 weeks of radiation. Carboplatin may be given as a substitution for cisplatin when cisplatin-related toxicities occur or when patients present with greater than grade 2 sensory or motor neuropathy, greater than 2 hearing loss, or less than 60 ml/min creatinine clearance.

SUMMARY:
This research is being done to try to reduce radiation side effects that happen with the standard radiation methods. Generally surgery, radiation therapy, and sometimes chemotherapy are standard treatment for people with squamous cell carcinoma of the oropharynx.

The study will look at giving a slightly smaller dose of radiation (de-intensification) to see if regularly expected late toxicities (two years after receiving treatment) can be reduced. This study will also try to see if the smaller dose of radiation is equally effective at treating the cancer and to see if it improves quality of life. Along with this radiation treatment plan some participants in this study will have surgery on their tumor and or receive chemotherapy (cisplatin or carboplatin). The possible surgery and or chemotherapy will be up to the participant's doctor.

Study participants will be tested for the Human Papillomavirus (HPV). This tissue test is required for this study. Some studies have suggested that HPV-related cancer is biologically and clinically different as compared to non-HPV-related cancer. Some studies have found that patients with HPV-related oropharynx cancer have a better response to treatment. This test will help researchers learn more about HPV-related cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven SCC of the oropharynx (tonsil, base of tongue, pharyngeal wall or palate).
* Tumor positive for infection with human papilloma virus (HPV) virus.
* T stage: 1, 2 or T3. Surgery of the primary tumor is limited to incisional or excisional biopsies (i.e tonsillectomy) even without macroscopic disease left. Positive resection margins and/or gross residual disease at the primary site are allowed.
* Any N stage, but resectable; lymph nodes in both sides of the neck are at risk of metastatic disease, according to clinical judgment, and require irradiation; pretreatment surgery in the neck in the forms of incisional/excisional biopsy or a multilevel neck dissection is allowed only if there is gross tumor left at the primary site.
* No other malignancy except for non-myelomatous skin cancer, early stage prostate cancer (T<2a and PSA<10 and GLS<7) or a carcinoma not of head and neck origin disease free for > 5 yrs.
* Cannot have distant metastasis (M0)
* ECOG performance status 0-1.
* Patient's nutritional and general physical condition must be considered compatible with the proposed radiotherapeutic treatment.
* Patient is judged to be mentally reliable to follow instructions and to keep appointments.
* Patient is on no other treatment for head and neck cancer.
* Signed study-specific informed consent prior to registration.

Exclusion Criteria:

* Evidence of distant metastases.
* Absence of macroscopic disease after upfront surgery
* Previous irradiation for head and neck tumor; concurrent chemotherapy other than the treatment per protocol; previous chemotherapy ≤ 3 months from start of RT.
* Active untreated infection.
* Major medical or psychiatric illness, which in the investigators' opinions would interfere with either completion of therapy and follow-up or with full and complete understanding of the risks and potential complications of the therapy.
* Prophylactic use of amifostine or pilocarpine is not allowed.
* Patients with greater than 1- pack years of smoking history and/or currently a smoker at the time of treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quon Harry, M.D., Principal Investigator — Johns Hopkins University; Arlene Forastiere, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from Johns Hopkins' Radiation/Medical Oncology clinics from 2010-2016.
Period: Overall Study
Arm/Group | Dose De-escalating Radiation Therapy With Chemotherapy
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dose De-escalating Radiation Therapy With Chemotherapy
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 59.3 [39.12 to 80.07]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white/caucasian | 56
  black/african american | 3
  hispanic/latino | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Free of Grade 3+ Late Toxicity
Description: The goal is to achieve a prevalence of < 15% grade 3+ late toxicity at 2 years; reported as percentage of patients who were free of grade 3+ adverse events (AEs) as measured by Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.0) between 6 months and 24 months. The outcome is reported as percentage of patients who were free of grade 3+ adverse events.
Time Frame: 2 years
Population: 5/60 patients did not have adverse event data captured for the period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose De-escalating Radiation Therapy With Chemotherapy
Number analyzed (Participants) | 55
percentage of participants | 86 [82 to 97]

2. Primary Outcome: Percentage of Patients With Locoregional Tumor Control
Description: Locoregional tumor control > 85 + or - 7% at 2 years; measured through progression-free survival (the time from assignment in a clinical trial to disease progression or death from any cause). Locoregional tumor control is reported as percentage of patients meeting this criteria.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose De-escalating Radiation Therapy With Chemotherapy
Number analyzed (Participants) | 60
percentage of participants | 92 [85 to 99]

3. Primary Outcome: Adverse Events and Their Cause
Description: To determine the nature and prevalence of side effects at different time intervals and describe their relationship to pretreatment function and local dose and treated volume.
Time Frame: Pretreatment, 3 months, then every 3 months for the first 2 years, then every 6 months for years 3-5
Population: Data was not collected to assess this outcome.
Arm/Group | Dose De-escalating Radiation Therapy With Chemotherapy
Number analyzed (Participants) | 0

4. Primary Outcome: Quality of Life Measured Through Patient-reported Outcome Measures on Assessments: M.D. Anderson Dysphagia Inventory (MDADI)
Description: Determine quality of life of surviving patients measured by patient reported outcomes:
  -MDADI-Self-administered assessment on patient swallowing ability. There are 19 questions specific to swallowing that study patients completed. Composite score is the average of the 19 questions. The scale is 20 (extremely low functioning) to 100 (high functioning).
  Composite score is reported.
Time Frame: Baseline, 6-8 weeks, 6 months, 1 year, 2 years, 3 years, 4-5 year visit
Population: Some patients did not respond to QoL assessment for the various time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose De-escalating Radiation Therapy With Chemotherapy
Number analyzed (Participants) | 48
score on a scale
  Baseline: number analyzed (Participants) | 45
  Baseline | 87.71 (13.72)
  6-8 week visit: number analyzed (Participants) | 40
  6-8 week visit | 77.75 (13.42)
  6 month visit: number analyzed (Participants) | 21
  6 month visit | 78.62 (13.45)
  1 year visit | 86.18 (11.86)
  2 year visit: number analyzed (Participants) | 43
  2 year visit | 87.64 (11.35)
  3 year visit: number analyzed (Participants) | 35
  3 year visit | 88.16 (9.68)
  4-5 year visit: number analyzed (Participants) | 44
  4-5 year visit | 89.48 (9.62)

5. Primary Outcome: Quality of Life Measured Through Patient-reported Outcome Measures on Assessments: MD Anderson Symptom Inventory-head and Neck Cancer (MDASI-HN)
Description: Determine quality of life of surviving patients measured by patient reported outcomes:
  MDASI-HN-Self-reported assessment. Measures symptom severity in previous day. Study patients answered 9 specific questions specific to head and neck cancer. Symptom severity scores, from 0 (not present) to 10 (worst possible). Composite score calculated average of individual scores.
  Mean module (head and neck) symptom severity is reported.
Time Frame: Baseline, 6-8 weeks, 1 year, 2 years, 3 years, 4-5 year visit
Population: Some patients did not respond to QoL assessment for the various time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose De-escalating Radiation Therapy With Chemotherapy
Number analyzed (Participants) | 56
score on a scale
  baseline: number analyzed (Participants) | 44
  baseline | 0.45 (0.6)
  6-8 week visit: number analyzed (Participants) | 52
  6-8 week visit | 4.17 (1.97)
  1 year visit | 1.06 (1.07)
  2 year visit | 0.98 (1.05)
  3 year visit: number analyzed (Participants) | 50
  3 year visit | 0.92 (1.02)
  4-5 year visit: number analyzed (Participants) | 43
  4-5 year visit | 0.9 (0.81)

6. Primary Outcome: Quality of Life Measured Through Patient-reported Outcome Measures on Assessments: Xerostomia Questionnaire (XQ)
Description: Determine quality of life of surviving patients measured by patient reported outcomes:
  XQ measures severity of radiation-induced xerostomia and patient reported quality of life. 8 question total:4 on dryness while eating/chewing, 4 on dryness when not eating/chewing. 0-10 (higher scores=severe dryness/discomfort). Composite Scores range from 0 (no xerostomia) -100 (highest level of xerostomia).
Time Frame: Baseline, 6-8 weeks, 1 year, 2 years, 3 years, 4-5 year visit
Population: Some patients did not respond to QoL assessment for the various time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose De-escalating Radiation Therapy With Chemotherapy
Number analyzed (Participants) | 56
score on a scale
  baseline: number analyzed (Participants) | 43
  baseline | 0.65 (0.89)
  6-8 week visit: number analyzed (Participants) | 52
  6-8 week visit | 6.23 (3.24)
  1 year visit | 3.27 (2.26)
  2 year visit | 2.96 (2.16)
  3 year visit: number analyzed (Participants) | 50
  3 year visit | 2.87 (1.96)
  4-5 year visit: number analyzed (Participants) | 44
  4-5 year visit | 2.67 (2.05)

ADVERSE EVENTS:
Time Frame: Up to 60 months after treatment
Description: Adverse events were collected using the CTCAE guide to assign category, term, and grade.
Arm/Group | Dose De-escalating Radiation Therapy With Chemotherapy
All-Cause Mortality (participants affected / at risk) | 1/60
Serious Adverse Events (participants affected / at risk) | 54/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose De-escalating Radiation Therapy With Chemotherapy (N=60)
abdominal pain (Gastrointestinal disorders) | 2 — Grade 3
akathisia (Nervous system disorders) | 1 — Grade 3
ANC decreased (Investigations) | 1 — Grade 3
Anemia (Blood and lymphatic system disorders) | 2 — Grade 3
anorexia (Metabolism and nutrition disorders) | 2 — Grade 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 — Grade 3
atrial fibrillation (Cardiac disorders) | 2 — Grade 3
back pain (Musculoskeletal and connective tissue disorders) | 1 — Grade 3
Chronic kidney disease (Renal and urinary disorders) | 1 — Grade 3
colonic obstruction (Gastrointestinal disorders) | 1 — Grade 3
constipation (Gastrointestinal disorders) | 1 — Grade 3
dehydration (Metabolism and nutrition disorders) | 6 — Grade 3
Dermatitis (Skin and subcutaneous tissue disorders) | 1 — Grade 3
diarrhea (Gastrointestinal disorders) | 1 — Grade 3
dysphagia (Gastrointestinal disorders) | 4 — Grade 3
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 — Grade 3
edema limbs (General disorders) | 1 — Grade 3
enterocolitis infectious (Infections and infestations) | 1 — Grade 3
Esophageal stricture (Gastrointestinal disorders) | 2 — Grade 3
fatigue (General disorders) | 5 — Grade 3
febrile neutropenia (Blood and lymphatic system disorders) | 4 — Grade 3
fever (General disorders) | 3 — Grade 3
flatulence (Gastrointestinal disorders) | 1 — Grade 3
general NOS: failure to thrive (General disorders) | 1 — Grade 3
hearing changes (Ear and labyrinth disorders) | 3 — Grade 3
Hyperglycemia (Metabolism and nutrition disorders) | 2 — Grade 3
Hyperkalemia (Metabolism and nutrition disorders) | 1 — Grade 3
Hypertension (Metabolism and nutrition disorders) | 1 — Grade 3
hypoglycemia (Metabolism and nutrition disorders) | 1 — Grade 3
Hypomagnesia (Metabolism and nutrition disorders) | 1 — Grade 3
Hyponatremia (Metabolism and nutrition disorders) | 2 — Grade 3
injury/procedure complication: bleeding at PEG site (Injury, poisoning and procedural complications) | 1 — Grade 3
injury/procedure complication: g-tube dysfunction (Injury, poisoning and procedural complications) | 1 — Grade 3
injury/procedure complication: PEG dysfunction (Injury, poisoning and procedural complications) | 2 — Grade 3
injury/procedure complication-NOS: admitted following left neck dissection (Injury, poisoning and procedural complications) | 1 — Grade 3
injury/procedure complication-NOS: PEG insertion (Injury, poisoning and procedural complications) | 1 — Grade 3
Leukocytosis (Blood and lymphatic system disorders) | 1 — Grade 3
lower GI hemorrhage (Gastrointestinal disorders) | 1 — Grade 3
lung infection (Respiratory, thoracic and mediastinal disorders) | 3 — Grade 3
lung metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Grade 3
lymphocytes decreased (Investigations) | 27 — Grade 3
Metastatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Grade 3
mucositis (Respiratory, thoracic and mediastinal disorders) | 28 — Grade 3
Mucous membrane (Respiratory, thoracic and mediastinal disorders) | 1 — Grade 3
Nausea (Gastrointestinal disorders) | 3 — Grade 3
oral pain (Gastrointestinal disorders) | 1 — Grade 3
pain (General disorders) | 3 — Grade 3
pain due to XRT (Injury, poisoning and procedural complications) | 5 — Grade 3
Pain NCI (General disorders) | 1 — Grade 3
pharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 — Grade 3
psych NOS (Psychiatric disorders) | 1 — Grade 3
restlessness (Psychiatric disorders) | 1 — Grade 3
saliva/salivary gland (Gastrointestinal disorders) | 11 — Grade 3
skin infection (Infections and infestations) | 1 — Grade 3
Subcutaneous tissue (Skin and subcutaneous tissue disorders) | 2 — Grade 3
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 — Grade 3
vascular access complication (Injury, poisoning and procedural complications) | 1 — Grade 3
venous thrombosis (Vascular disorders) | 1 — Grade 3
Voice changes (Respiratory, thoracic and mediastinal disorders) | 1 — Grade 3
Vomiting (Gastrointestinal disorders) | 3 — Grade 3
WBC Decreased (Investigations) | 2 — Grade 3
Xerostomia (Gastrointestinal disorders) | 1 — Grade 3
lymphocytes decreased (Investigations) | 23 — Grade 4
Neutrophils decreased (Investigations) | 1 — Grade 4
pain (Injury, poisoning and procedural complications) | 1 — Grade 4
PsychNOS: mood disorder (Psychiatric disorders) | 1 — Grade 4
WBC Decreased (Investigations) | 4 — Grade 4
injury to carotid artery (Injury, poisoning and procedural complications) | 1 — Grade 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose De-escalating Radiation Therapy With Chemotherapy (N=60)
ALT increased (Investigations) | 22 — Grade 1
anemia (Blood and lymphatic system disorders) | 49 — Grade 1
aspiration (Respiratory, thoracic and mediastinal disorders) | 17 — Grade 1
AST increased (Investigations) | 6 — Grade 1
bilirubin increased (Investigations) | 5 — Grade 1
cough (Respiratory, thoracic and mediastinal disorders) | 20 — Grade 1
creatinine increased (Investigations) | 12 — Grade 1
dehydration (Metabolism and nutrition disorders) | 11 — Grade 1
dermal caries (Gastrointestinal disorders) | 10 — Grade 1
dermatitis (Skin and subcutaneous tissue disorders) | 9 — Grade 1
dysgeusia (Nervous system disorders) | 16 — Grade 1
dysphagia (Gastrointestinal disorders) | 35 — Grade 1
esophageal stenosis (Gastrointestinal disorders) | 8 — Grade 1
esophagus/RTOG (Gastrointestinal disorders) | 3 — Grade 1
fatigue (General disorders) | 28 — Grade 1
hearing changes (Ear and labyrinth disorders) | 4 — Grade 1
hyperglycemia (Metabolism and nutrition disorders) | 45 — Grade 1
hyperkalemia (Metabolism and nutrition disorders) | 8 — Grade 1
hypoalbuminemia (Metabolism and nutrition disorders) | 3 — Grade 1
hypocalcemia (Metabolism and nutrition disorders) | 6 — Grade 1
hypomagnesia (Metabolism and nutrition disorders) | 5 — Grade 1
hyponatremia (Metabolism and nutrition disorders) | 19 — Grade 1
larynx/RTOG (Respiratory, thoracic and mediastinal disorders) | 15 — Grade 1
mucositis (Respiratory, thoracic and mediastinal disorders) | 11 — Grade 1
mucous membrane/RTOG (Respiratory, thoracic and mediastinal disorders) | 27 — Grade 1
nausea (Gastrointestinal disorders) | 33 — Grade 1
pain due to XRT (Injury, poisoning and procedural complications) | 16 — Grade 1
platelets/count decreased (Investigations) | 29 — Grade 1
saliva/salivary gland (Gastrointestinal disorders) | 6 — Grade 1
skin acute (Skin and subcutaneous tissue disorders) | 12 — Grade 1
skin acute (Skin and subcutaneous tissue disorders) | 5 — Grade 1
skin late (Skin and subcutaneous tissue disorders) | 25 — Grade 1
subcutaneous tissue/RTOG (Skin and subcutaneous tissue disorders) | 34 — Grade 1
tinnitus (Ear and labyrinth disorders) | 36 — Grade 1
trismus (Musculoskeletal and connective tissue disorders) | 13 — Grade 1
voice changes/alteration (Respiratory, thoracic and mediastinal disorders) | 38 — Grade 1
vomiting (Gastrointestinal disorders) | 13 — Grade 1
watery eye (Eye disorders) | 3 — Grade 1
WBC decreased (Investigations) | 30 — Grade 1
weight loss (Investigations) | 26 — Grade 1
xerostomia (Gastrointestinal disorders) | 4 — Grade 1
anemia (Blood and lymphatic system disorders) | 7 — Grade 2
anorexia (Metabolism and nutrition disorders) | 6 — Grade 2
dehydration (Metabolism and nutrition disorders) | 6 — Grade 2
dermatitis (Skin and subcutaneous tissue disorders) | 28 — Grade 2
dysgeusia (Nervous system disorders) | 41 — Grade 2
dysphagia (Gastrointestinal disorders) | 14 — Grade 2
esophagitis (Gastrointestinal disorders) | 5 — Grade 2
esophagus/RTOC (Gastrointestinal disorders) | 8 — Grade 2
fatigue (General disorders) | 22 — Grade 2
hearing changes/impairment (Ear and labyrinth disorders) | 5 — Grade 2
hyperglycemia (Metabolism and nutrition disorders) | 9 — Grade 2
hypomagnesia (Metabolism and nutrition disorders) | 3 — Grade 2
larynx/RTOG (Respiratory, thoracic and mediastinal disorders) | 8 — Grade 2
lymphocytes decreased (Investigations) | 6 — Grade 2
mucositis (Respiratory, thoracic and mediastinal disorders) | 21 — Grade 2
mucous membrane/RTOG (Respiratory, thoracic and mediastinal disorders) | 11 — Grade 2
nausea (Gastrointestinal disorders) | 19 — Grade 2
neuralgia (Nervous system disorders) | 3 — Grade 2
neutrophil count decreased (Investigations) | 5 — Grade 2
pain due to XRT (Injury, poisoning and procedural complications) | 32 — Grade 2
salivary gland (Gastrointestinal disorders) | 48 — Grade 2
skin acute (Skin and subcutaneous tissue disorders) | 43 — Grade 2
skin late (Skin and subcutaneous tissue disorders) | 5 — Grade 2
subcutaneous tissue (Skin and subcutaneous tissue disorders) | 13 — Grade 2
tinnitus (Ear and labyrinth disorders) | 7 — Grade 2
voice changes (Respiratory, thoracic and mediastinal disorders) | 7 — Grade 2
vomiting (Gastrointestinal disorders) | 4 — Grade 2
WBC decreased (Investigations) | 15 — Grade 2
weight loss (Investigations) | 13 — Grade 2
xerostomia (Gastrointestinal disorders) | 53 — Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT01088802/Prot_SAP_000.pdf